CLINICAL TRIAL: NCT06111794
Title: The REACH Intervention for Caregivers of Veterans and Service Members With TBI: Efficacy and Implementation Planning Across the VA Polytrauma System of Care
Brief Title: The REACH Intervention for Caregivers of Veterans and Service Members With TBI
Acronym: REACH TBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: James A. Haley Veterans Administration Hospital (U.S. Federal Agency); Virginia Commonwealth University (Other); University of Utah (Other); University of Tennessee (Other)
Responsible Party: Principal Investigator, Paul B. Perrin, Professor of Data Science and Psychology, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CDMRP-TP220091
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Traumatic Brain Injury; Caregiver
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: This study uses a treatment/waitlist-control crossover repeated-measures design.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REACH TBI (Experimental): Participants will receive the REACH TBI psychoeducational intervention.
  Interventions: Other: REACH TBI
- Waitlist Control (Active Comparator): Participants will receive the REACH TBI psychoeducational intervention.
  Interventions: Other: REACH TBI

INTERVENTIONS:
Other: REACH TBI — Resources for Enhancing All Caregivers' Health - Traumatic Brain Injury (REACH TBI) is a six-session, telephone intervention for Caregivers of Veterans and Services Members with TBI. The intervention focuses on problem solving training, stress management, and psychoeducation. Trained Program Coaches will deliver the REACH TBI intervention by meeting one-on-one via telephone with participants.

SUMMARY:
This randomized waitlist control trial will evaluate the effects of a psychoeducational intervention called Resources for Enhancing All Caregivers' Health - Traumatic Brain Injury (REACH TBI) to decrease caregiver strain (primary outcome) and improve caregiver self-efficacy, anxiety, depression, and health care frustrations (secondary outcomes). This study will modify and adapt an award-winning caregiver intervention, Resources for Enhancing All Caregivers Health in the Department of Veterans Affairs (REACH VA), to support the needs of Caregivers of Veterans and Service Members with TBI.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, the participant must:

* identify as a primary caregiver for a V/SM who sustained a TBI at least 6 months prior;
* identify as a primary caregiver who has provided care for a V/SM with TBI for at least 6 months;
* provide some level of daily supervision or assistance with either a physical, cognitive, or behavioral issue they think is likely related to TBI;
* believe that at least half of their caregiving responsibilities are likely related to TBI rather than another health condition(s); and
* endorse a score of at least high burden (a score of 8 or higher) on the Zarit Burden Inventory-4.

Exclusion Criteria:

* no telephone;
* current diagnosis of schizophrenia or other major mental illness;
* auditory impairment that would make telephone use difficult; or
* the caregiver believes that more than half of their caregiving for the V/SM is for issues related to another health condition(s) rather than TBI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
TBI-CareQOL Caregiver Strain - Short Form 6a | Baseline; 3 months (post-intervention); 6 month follow-up
  It assesses caregiver strain in caregivers of individuals with TBI. Values range from 6-30, with higher scores indicating greater strain/worse outcome.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System Emotional Distress - Depression - Short Form 4a | Baseline; 3 months (post-intervention); 6 month follow-up
  It assesses caregiver depression. Values range from 8-40, with higher scores indicating greater depression/worse outcome.
Patient-Reported Outcomes Measurement Information System Emotional Distress - Anxiety - Short Form 4a | Baseline; 3 months (post-intervention); 6 month follow-up
  It assesses caregiver anxiety. Values range from 7-35, with higher scores indicating greater anxiety/worse outcome.
Patient-Reported Outcomes Measurement Information System - General Self-Efficacy | Baseline; 3 months (post-intervention); 6 month follow-up
  It assesses caregiver self-efficacy. Values from range 10-50, with higher scores indicating greater self-efficacy/better outcome.
TBI-CareQOL Health Care Frustration - Self - Short Form 6a | Baseline; 3 months (post-intervention); 6 month follow-up
  It assesses frustrations a TBI caregiver has had with health care services. Values range from 6-30, with higher scores indicating greater frustration with services received/worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampa VA Medical Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data are available to other researchers via FITBIR.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the end of data collection and cleaning and will be available for a period of at least 5 years.